CLINICAL TRIAL: NCT05420051
Title: A Novel Psychological-behavioral Intervention to Promote Physical Activity in Type 2 Diabetes
Brief Title: Boosting Emotional Well-being and Happiness in Outpatients Living With Diabetes
Acronym: BEHOLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P000780
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Psychology, Positive; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology + Motivational Interviewing (Experimental): Each week, participants in the PP-MI intervention group will complete a PP activity and work towards a physical activity goal, then complete a phone session with a study trainer. Each phone session will include PP and goal setting portions. In the PP portion, the study trainer will (a) review the week's PP exercise, (b) discuss the rationale of the next week's PP exercise through a guided review of the PP-MI manual, and (c) assign the next week's PP exercise. In the goal-setting portion, the trainer will (a) review the participant's physical activity goal from the prior week, (b) discuss techniques for improving physical activity (e.g. tracking activity), and (c) help the participant to set a physical activity goal for the next week. Participants also will receive supplemental text messages throughout the 8 weeks of the intervention and during the initial follow-up period (Week 9-16).
  Interventions: Behavioral: Positive Psychology + Motivational Interviewing
- Motivational Interviewing (Active Comparator): Each week, participants in the MI-alone group will complete an activity related to a health behavior (e.g., thinking about the pros and cons of changing the behavior), then complete a phone session with a study trainer. During the phone session, the trainer will (a) review the prior week's topic, (b) discuss techniques for improving adherence to health behaviors (e.g. tracking activity), and (c) problem-solve barriers and encourage the use of resources. Participants also will receive supplemental text messages throughout the 8 weeks of the intervention and during the initial follow-up period (Week 9-16).
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Positive Psychology + Motivational Interviewing — The 8-week PP-MI intervention focuses on enhancing well-being (through PP) and increasing physical activity (through MI). Each week, participants will complete a PP activity and work towards a physical activity goal, then complete a phone session with a study trainer. The PP portion of the program will focus on the cultivation of well-being through the performance of easy-to complete activities (e.g., using a strength in a new way) and review of the positive feelings they generate. The MI portion of the program will focus on assisting participants to improve physical activity levels, resolve ambivalence to behavior change, set realistic physical activity goals, problem-solve barriers, and identify resources to complete behavior change. Finally, participants will receive twice weekly text messages (for 16 weeks) to encourage completion of PP activities and engagement in physical activity.
  Arms: Positive Psychology + Motivational Interviewing
Behavioral: Motivational Interviewing — The 8-week MI-alone intervention focuses on providing education and enhancing motivation to engage in health behaviors (through MI). Each week, participants will complete an activity related to a health behavior (e.g., consider the pros and cons of behavior change, set a health behavior goal), then complete a phone session with a study trainer. This program will focus on assisting participants to improve health behavior adherence (including physical activity), resolve ambivalence to behavior change, set realistic health behavior goals, problem-solve barriers, and identify resources to complete behavior change. Additional time in MI-alone phone sessions will be spent on review of core MI skills, problem-solving of barriers, and discussion of resources. Finally, participants will receive twice weekly text messages (for 16 weeks) to encourage engagement in health behaviors.
  Arms: Motivational Interviewing

SUMMARY:
The focus of this study is to test the efficacy of an 8-week, remotely delivered, positive-psychology-motivational interviewing (PP-MI) intervention, with additional twice weekly text messages for a total of 16 weeks (with interactive, algorithm-driven, goal-focused text messages in the final 8 weeks), compared to MI-alone, in a randomized trial of 280 individuals with type 2 diabetes and low baseline physical activity.

DETAILED DESCRIPTION:
The investigators are proposing a study that will focus on testing the efficacy of a PP-MI intervention, with additional twice text messages for a total of 16 weeks (with interactive, algorithm-driven, goal-focused text messages in the final 8 weeks) in individuals with type 2 diabetes. The investigators will enroll 280 type 2 diabetes patients, who will take part in either an 8-week intervention (with 16 weeks of supplemental text messages) or an attention-matched, MI-alone condition.

In this project, the investigators hope to do the following:

1. Examine the efficacy of an 8-week, phone-delivered PP-MI intervention for individuals with type 2 diabetes on physical activity-related outcomes, as compared to the MI-alone condition.
2. Assess PP-MI's impact on psychological measures (e.g., positive affect [key secondary outcome]), diabetes self-care, function, glycemic control, and cardiometabolic risk, compared to MI alone.
3. Examine causal mediation of PP-MI's effects on MVPA at 16 weeks by positive affect (primary hypothesized mediator) and other psychological/cognitive variables across our theoretical model.

Participants will be adult outpatients with type 2 diabetes. They will attend an in-person visit to provide informed consent and complete baseline outcome measures, then will wear an accelerometer to monitor their physical activity for one week to obtain information about baseline activity levels. Upon confirmation of low moderate to vigorous physical activity, participants will be randomized to receive the PP-MI intervention or the MI-alone intervention.

Participants in both groups will be provided a treatment manual, an activity tracker, and other treatment materials. The intervention will be introduced, and the first exercise will be assigned.

Participants will complete eight weekly phone sessions with a study trainer. The phone sessions primarily will include a review of the prior week's session content and a discussion of the rationale and assignment of the next week's exercise/assignment.

Participants will receive twice weekly text messages throughout the intervention (Weeks 1-8) and initial follow-up period (Weeks 9-16). In the PP-MI condition, these messages will focus on the PP activity and physical activity, while those in the MI-alone condition will focus on physical activity and other health behaviors. During Weeks 9-16, participants in the PP-MI condition will engage with twice weekly, automated, interactive text messages related to PP and physical activity, while those in the MI-alone condition will receive fixed text messages related to engagement in health behaviors.

At Weeks 8, 16, 24, and 52, participants will complete follow-up visits. One week prior to these visits, participants will be mailed an accelerometer and will wear it until their study visit. During these study visits, participants will complete outcome assessments and have a blood sample taken.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes
* Low physical activity (<150 minutes/week of moderate to vigorous physical activity)

Exclusion Criteria:

* Cognitive deficits impeding a participant's ability to provide informed consent or participate
* Medical conditions likely to lead to death within 6 months.
* Pre-existing coronary artery disease
* Moderate-severe depression (Patient Health Questionnaire-9 [PHQ-9] score ≥15)
* Use of non-basal insulin
* Inability to participate in physical activity due to another medical condition
* Inability to receive text messages
* Inability to read, write, or speak in English
* Current participation in another intervention or program that has been designed to promote well-being or physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Moderate to Vigorous Physical Activity (MVPA) at 16 weeks | Measured for 7 days at baseline and 16 weeks
  MVPA will be measured via an accelerometer and recorded in mean minutes/day.

SECONDARY OUTCOMES:
Change from Baseline Overall Activity at 16 weeks | Measured for 7 days at baseline and 16 weeks
  Overall activity will be measured via an accelerometer and recorded in mean steps/day.
Change from Baseline in positive affect (Positive and Negative Affect Schedule [PANAS] positive affect items) at 16 weeks | Baseline, 16 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.

OTHER OUTCOMES:
Change from Baseline Moderate to Vigorous Physical Activity (MVPA) at 8, 24, and 52 weeks | Measured for 7 days at baseline, 8 weeks, 24, weeks, and 52 weeks
  MVPA will be measured via an accelerometer and recorded in mean minutes/day.
Change from Baseline Overall Activity at 8, 24, and 52 weeks | Measured for 7 days at baseline, 8 weeks, 24, weeks, and 52 weeks
  Overall activity will be measured via an accelerometer and recorded in mean steps/day.
Change from Baseline in positive affect (Positive and Negative Affect Schedule [PANAS] positive affect items) at 8, 24, and 52 weeks | Baseline, 8 weeks, 24 weeks, 52 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.
Change in optimism (Life Orientation Test - Revised [LOT-R]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of dispositional optimism.
Change in depressive symptoms (Patient Health Questionnaire [PHQ-9]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  The Patient Health Questionnaire-9 (PHQ-9) will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-27). Higher scores indicate higher levels of depression.
Change in anxiety (Hospital Anxiety and Depression Scale - anxiety subscale [HADS-A]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale will be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety.
Change in locus of control (Form C of the Multidimensional Health Locus of Control scale [MHLC Form C]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Locus of control will be measured using the 18-item Multidimensional Health Locus of Control scale [MHLC Form C]. Scores on this scale range from 6-36, with higher scores indicating greater internal health locus of control.
Change in perceived social support (Multidimensional Scale of Perceived Social Support [MSPSS]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  The MSPSS is a 12-item scale designed to measure perceived social support from three sources: Family, Friends, and a Significant Other. Scores on this scale range from 0-84, with higher scores indicating greater perceived social support.
Change in exercise-related self-efficacy (Self-efficacy for Exercise Scale [SEE]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  The Self-efficacy for Exercise Scale will be used to measure exercise self-efficacy. This is a 9-item scale used to assess an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 20+ minutes per session in the future. Scores on this scale range from 0-90, with higher scores indicating greater self-efficacy for exercise.
Change in physical function (PROMIS 20-item Physical Function Short Form [PF-20]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  The PROMIS 20-item short form (PF-20) will be used to assess physical function. Scores on this scale range from 20-100, with higher scores indicating greater physical function.
Change in mental health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12] mental component score) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  The SF-12 mental component score will be used to assess mental health-related quality of life (Range: 0-100). Higher scores indicate higher levels of mental health-related quality of life.
Change in physical health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12] physical component score) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  The SF-12 physical component score will be used to assess physical health-related quality of life (Range: 0-100). Higher scores indicate higher levels of physical health-related quality of life.
Change in adherence to a diabetes diet (General diet items of the Summary of Diabetes Self-Care Activities [SDSCA]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Measured by the general diet items of the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate greater adherence.
Change in adherence to fruits, vegetables, and low fat foods (Specific diet items of the Summary of Diabetes Self-Care Activities [SDSCA]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Measured by the specific diet items of the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate greater adherence.
Change in exercise (Exercise items of the Summary of Diabetes Self-Care Activities [SDSCA]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Measured by the exercise items of the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate more exercise.
Change in frequency of blood glucose testing (Blood glucose testing items of the Summary of Diabetes Self-Care Activities [SDSCA]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Measured by the blood glucose testing items of the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate more frequent blood glucose testing.
Change in foot care (Foot care items of the Summary of Diabetes Self-Care Activities [SDSCA]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Measured by the foot care items of the Summary of Diabetes Self-Care Activities (SDSCA), a well-validated measure of diabetes self-management that is associated with clinical outcomes (Range: 0-7). Higher scores indicate more frequent foot care.
Change in self-reported MVPA (International Physical Activity Questionnaire [IPAQ]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assesses the types of intensity of physical activity that people do as part of their daily lives. Moderate and vigorous intensity activities will be converted to multiples of resting energy expenditure (MET) minutes per week.
Change in self-reported sedentary time (International Physical Activity Questionnaire [IPAQ]) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Measured by the self-report International Physical Activity Questionnaire (IPAQ). Measured in hours per day.
Change in weight (kilograms) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Weight will be measured during study visits.
Change in body mass index (kilograms per square meter) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Height and weight will be measured during study visits.
Change in blood pressure (millimeters of mercury) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Blood pressure (diastolic and systolic) will be measured by trained nurses using a standardized protocol.
Change in hemoglobin A1C (%) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Blood samples will be obtained at study visits.
Change in low density lipoprotein (LDL) and high density lipoprotein (HDL) cholesterol (milligrams per deciliter) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Blood samples will be obtained at study visits.
Change in triglycerides (milligrams per deciliter) | Baseline, 8 weeks, 16 weeks, 24 weeks, 52 weeks
  Blood samples will be obtained at study visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
To promote sharing of study data with other researchers, we will create a deidentified study dataset. We will include both item-level and summary scores for each scale and will include data from the baseline, 8-week, 16-week, 24-week, and 52-week time points.
Supporting Information: Study Protocol, SAP
Time Frame: This information will be shared prior to the end of the study funding period.
Access Criteria: Investigators who are interested in obtaining access to this information will be asked to submit a request to the principal investigator outlining the proposed use of the data and would need to agree to certain conditions (e.g., not attempting to identify individual participants, destroying data once the use of the data is complete) prior to obtaining access.